CLINICAL TRIAL: NCT00974220
Title: Effect of Inhaled Nebulized Fentanyl on Exertional Dyspnea and Exercise Tolerance in Patients With Moderate-to-severe COPD
Brief Title: Effect of Inhaled Fentanyl on Dyspnea and Exercise Tolerance in Chronic Obstructive Pulmonary Disease (COPD)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Queen's University (Other)
Responsible Party: Principal Investigator, Dr. Denis O'Donnell, Principal Investigator, Queen's University
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DSS16327
Record Dates: First submitted 2009-09-09; First posted 2009-09-10 (Estimated); Results first posted 2015-12-30 (Estimated); Last update posted 2019-07-12 (Actual); Status verified 2019-07

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: inhaled fentanyl; dyspnea; exercise; COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Dyspnea; Motor Activity | interventions — Fentanyl; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- placebo (Placebo Comparator): nebulized 0.9% saline placebo
  Interventions: Drug: normal saline (placebo)
- fentanyl (Experimental): nebulized fentanyl citrate (50 mcg)
  Interventions: Drug: fentanyl

INTERVENTIONS:
Drug: fentanyl — single dose, 50 mcg of nebulized fentanyl citrate
  Arms: fentanyl
Drug: normal saline (placebo) — single dose, 0.9% saline solution
  Arms: placebo

SUMMARY:
Breathing discomfort (dyspnea) and activity limitation are dominant symptoms of chronic obstructive pulmonary disease (COPD) and contribute to poor health-related quality of life in this population. Several small, uncontrolled studies and published case reports have provided evidence that inhaled fentanyl, a powerful pain relieving (opioid) medication, may be used to effectively reduce breathing discomfort in patients with advanced disease. However, the mechanisms of this improvement remain unclear. Therefore, the investigators plan to conduct the first randomized, double-blind, placebo-controlled, crossover study designed to explore the possible mechanisms of action of inhaled fentanyl on activity-related dyspnea and exercise performance in patients with advanced COPD.

ELIGIBILITY:
Inclusion Criteria:

* Post-bronchodilator forced expiratory volume in 1 sec (FEV1) 30-79% predicted, FEV1/forced vital capacity (FVC) ratio <70%;
* Clinically stable as defined by no changes in medication dosage or frequency of administration with no exacerbations or hospital admissions in the preceding 6 weeks;
* A cigarette smoking history ≥20 pack-years;
* Significant chronic activity-related dyspnea as defined by a Baseline Dyspnea Index focal score ≤ 6;
* Body mass index (BMI) between 18.5 and 30.0 kg/m2;
* Able to perform all study procedures and provide/sign informed consent.

Exclusion Criteria:

* A diffusing capacity of the lung for carbon monoxide (DLCO) <40 %predicted;
* Presence of active cardiopulmonary disease other than COPD that could contribute to dyspnea and exercise limitation;
* Clinical diagnosis of sleep disordered breathing;
* A history/clinical evidence of asthma, atopy and/or nasal polyps;
* History of allergy or adverse reaction to fentanyl;
* Presence of important contraindications to clinical exercise testing, including inability to exercise because of neuromuscular or musculoskeletal disease(s);
* Use of daytime oxygen or exercise-induced arterial oxygen desaturation to <80% on room air;
* Use of antidepressant drugs (i.e., monoamine oxidase inhibitors, serotonin reuptake inhibitors) in previous 2 weeks;
* Use of opioid or pain relieving drugs (e.g., morphine, fentanyl, oxycodone, hydromorphone, methadone, levorphanol, codeine, hydrocodone, meperidine) in previous 4 weeks.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2010-01; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Denis E O'Donnell, MD, FRCPC, Principal Investigator — Queen's University and Kingston General Hospital; Deborah Dudgeon, MD, FRCPC, Principal Investigator — Queen's University and Kingston General Hospital
Locations (1):
- Respiratory Investigation Unit, Kingston General Hospital, Kingston, Ontario, Canada

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment took place between February and October 2010. Subjects were recruited from respiratory outpatient clinics and from a database of subjects who had previously taken part in research studies in COPD.
Pre-assignment Details: No enrolled subjects were excluded prior to group assignment.
  7 subjects were assigned a treatment order of fentanyl-placebo (2 were withdrawn after period 1) and 9 subjects were assigned a treatment order of placebo-fentanyl (2 were withdrawn after period 1). Therefore, there was complete data from 12 subjects.
Groups:
- Placebo - Fentanyl (Order): nebulized 0.9% saline placebo in period 1, nebulized fentanyl citrate 50mcg in period 2
- Fentanyl - Placebo (Order): nebulized fentanyl citrate (50 mcg) in period 1, nebulized 0.9% saline placebo in period 2
Period: Treatment Period 1
Arm/Group | Placebo - Fentanyl (Order) | Fentanyl - Placebo (Order)
Started | 9 | 7
Completed | 7 | 5
Not Completed | 2 | 2
Not completed — Adverse Event | 2 | 1
Not completed — noncompliant subjects | 0 | 1
Period: Treatment Period 2
Arm/Group | Placebo - Fentanyl (Order) | Fentanyl - Placebo (Order)
Started | 7 | 5
Completed | 7 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Placebo - Fentanyl (Order): nebulized saline placebo in period 1, nebulized fentanyl citrate in period 2.
- Fentanyl - Placebo (Order): nebulized fentanyl citrate in period 1, nebulized saline placebo in period 2.
- Total: Total of all reporting groups
Arm/Group | Placebo - Fentanyl (Order) | Fentanyl - Placebo (Order) | Total
Number analyzed (Participants) | 9 | 7 | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 69 (8) | 66 (10) | 68 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 7
  Male | 6 | 3 | 9
Region of Enrollment [Number; unit: participants]
  Canada | 9 | 7 | 16

OUTCOME MEASURES:

1. Primary Outcome: Dyspnea Intensity Measured by the 10-point Borg Scale During Cycle Exercise
Description: The 10-point Borg scale ranges from 0 "nothing at all" to 10 "maximal/extremely strong" and was used to rate the intensity of dyspnea during exercise; therefore, a decrease in this rating signifies an improvement. Dyspnea intensity was assessed at the highest equivalent standardized time achieved in both post-treatment constant work rate cycle exercise tests.
Time Frame: 10-minutes post-treatment
Population: Subjects who completed both treatment arms of the crossover study were included in the primary analysis.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Fentanyl
Number analyzed (Participants) | 12 | 12
units on a scale | 2.6 (0.5) | 2.0 (0.5)

2. Secondary Outcome: Cycle Exercise Endurance Time
Description: Constant workrate cycle endurance during tests at 75% of the peak incremental workrate
Time Frame: 10-minutes post-treatment
Population: Subjects completing both treatment arms were included in this analysis
Measure: Mean (Standard Error); unit: minutes
Arm/Group | Placebo | Fentanyl
Number analyzed (Participants) | 12 | 12
minutes | 6.04 (0.56) | 7.34 (0.70)

ADVERSE EVENTS:
Time Frame: During visit, with appropriate follow-up to resolution of adverse event
Arm/Group | Placebo | Fentanyl
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/16
Other Adverse Events (participants affected / at risk) | 2/16 | 1/16
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=16) | Fentanyl (N=16)
lightheadedness, dizziness and mild nausea (Nervous system disorders) | 1 (1) | 1 (1) — Lightheadedness, dizziness and mild nausea was experienced during and immediately after nebulization of the study medication. Symptoms quickly resolved but resulted in discontinuation from the study.
severe dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — Severe dyspnea was experienced during the nebulization of study medication. This resolved quickly after discontinuing nebulization but resulted in withdrawal from the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No